CLINICAL TRIAL: NCT06487377
Title: A Clinical Study of IX001 TCR-T In the Treatment of Advanced Pancreatic Cancer and Colorectal Cancer Induced by KRAS Mutations
Brief Title: IX001 TCR-T In the Treatment of Advanced Pancreatic Cancer and Colorectal Cancer Induced by KRAS Mutations
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pudong Hospital (Other)
Collaborators: ImmuXell Biotech Ltd. (Unknown)
Responsible Party: Principal Investigator, Minghua Yu, Dr, Chief physician, Shanghai Pudong Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT003
Record Dates: First submitted 2024-06-07; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Cancer; Colorectal Cancer
Keywords: KRAS-G12V or G12D
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IX001 TCR-T cells (Experimental): IX001 TCR-T cells targeted for KRAS mutation
  Interventions: Biological: IX001 TCR-T cells

INTERVENTIONS:
Biological: IX001 TCR-T cells — IX001 TCR-T cell injection will be administered intravenously after lymphodepletion.

SUMMARY:
This is a single-arm, single-center, open-label clinical study aimed at evaluating the safety and efficacy of IX001 TCR-T (T cell receptor-engineered T-Cell) injection in patients with advanced pancreatic cancer and colorectal cancer induced by KRAS (Kirsten Rat Sarcoma Viral Oncogene) mutations. A total of 6-18 evaluable patients are planned to be enrolled. The study will include 4 dose groups, using a '3+3' dose escalation design.

DETAILED DESCRIPTION:
Patients who sign the informed consent form will undergo screening based on inclusion/exclusion criteria. Eligible patients will be enrolled sequentially into dose group 1, dose group -1 or dose group 2, and dose group 3. The procedure of this study is as follows:

(I) The collected peripheral blood mononuclear cells (PBMCs) will be transported to the production workshop for the preparation of IX001. After confirming that IX001 is proved qualified, the investigator will decide whether to start pre-conditioning 5 days before IX001 infusion.

(II) TCR-T cells will be administered via intravenous infusion, and the cell infusion dose will be determined according to the requirements of dose escalation.

(III) Following TCR-T cell infusion, recombinant human interleukin-2 (IL-2) will be continuously injected to assist TCR-T cell growth.

(IV) After TCR-T cell infusion and IL-2 injection are completed, safety and efficacy follow-up visits will be conducted with the subjects until week 96 or until the subject prematurely withdraws from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of an informed consent form (ICF);
2. Males or females, aged 18-70 years (inclusive);
3. Pathologically diagnosed with advanced pancreatic cancer or colorectal cancer, having failed or intolerant to at least two lines of standard of care, including metastatic tumors (having received conventional chemotherapy), recurrent tumors (having undergone surgery and adjuvant chemotherapy in the past), or locally advanced tumors with disease progression after neoadjuvant treatment;
4. At least one measurable lesion (according to RECIST1.1[The Response Evaluation Criteria In Solid Tumors] criteria);
5. Patients with tumor tissue or peripheral blood testing positive for KRAS-G12V or G12D mutations and expression of matching HLA-A*11, C*01:02, or C*08:02 subtypes;
6. ECOG (Eastern Cooperative Oncology Group)≤2;
7. Life expectancy ≥3 months;
8. Absolute neutrophil count ≥1×10E9/L;
9. Platelet count ≥50×10E9/L, hemoglobin>90g/dL;
10. Absolute lymphocyte count ≥0.5×10E9/L;
11. Adequate functional reserve of organs:

    1. Aspartate aminotransferase ≤2.5×ULN (upper limit of normal);
    2. Aspartate transaminase ≤2.5×ULN;
    3. Creatinine clearance ≥60mL/min;
    4. Total serum bilirubin ≤1.5×UNL;
    5. The subject has left ventricular ejection fraction (LVEF) ≥ 50% and no clinically significant pericardial effusion diagnosed by echocardiography;
    6. No clinically significant electrocardiographic abnormality;
    7. Basic oxygen saturation is >92% under the indoor natural air environment.
12. Women of childbearing age must be negative for blood HCG (Human Chorionic Gonadotropin) pregnancy test (by immunofluorescence method) at screening and baseline periods, and agree to use effective contraception for at least 1 year after infusion; and male subjects whose partners are women of childbearing age must agree to use effective barrier contraception methods and avoid sperm donation for at least 1 year after infusion. Contraception must include one highly effective and one additional effective (barrier) method, initiated from screening until at least 1 year after IX001 infusion or until two consecutive flow cytometry tests show the absence of TCR-T cells (whichever occurs later).

Exclusion Criteria:

1. Other malignancies (except non-melanoma skin cancer with the disease-free survival of more than 5 years and cervical carcinoma in situ, bladder cancer, or breast cancer);
2. A history of mental disorders, which may affect compliance with this protocol or lead to failure in signing the ICF;
3. Poorly controlled hypertension with drug (systolic blood pressure >160 mmHg and/or diastolic blood pressure >90 mmHg) or occurrence of grade III-IV heart failure or myocardial infarction, cardiac angioplasty or stent placement, unstable angina pectoris, or other clinically significant heart diseases within one year prior to signing the ICF; QTc interval >450 ms for males or QTc interval >470 ms for females during screening (QTc interval calculated using the Fridericia formula);
4. Presence of any indwelling catheter or drainage tube (e.g., percutaneous nephrostomy tube, indwelling catheter, bile drainage tube or pleural/peritoneal/pericardial catheter), except any dedicated central venous catheter;
5. A history of or any central nervous system disorders, such as epileptic seizure, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving the central nervous system;
6. A positive result obtained in any of the following virological tests:

   1. Antibody to human immunodeficiency virus (HIV antibody);
   2. Hepatitis C virus antibody (HCV antibody), with a positive result for hepatitis C virus ribonucleic acid (HCV RNA);
   3. Positive for hepatitis B surface antigen (HBsAg); or positive for hepatitis B core antibody (HBcAb) and positive for hepatitis B virus deoxyribonucleic acid (HBV DNA) copies;
   4. Treponema pallidum antibody (TP antibody); patients may be enrolled after additional examinations are performed to exclude active syphilis where necessary;
7. Fungal, bacterial, viral or other infections or suspected fungal, bacterial, viral or other infections that cannot be controlled or require intravenous administration;
8. Significant tendency for bleeding, such as active gastrointestinal bleeding, coagulation disorders;
9. Patients with a history of severe allergy or allergic constitution;
10. A history of autoimmune diseases (e.g., Crohn's disease, rheumatoid arthritis and systemic lupus erythematosus) requiring systemic immunosuppressive/systemic disease-modulating drugs in the past 2 years;
11. Interstitial lung disease (such as pneumonia, pulmonary fibrosis), or a history of clinically significant respiratory system diseases during screening;
12. History of organ transplantation;
13. Use of granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 2 weeks prior to leukapheresis;
14. Receipt of gene therapy or other cell therapies with the same target within the past 6 months;
15. Participation in any other clinical trial within 4 weeks prior to signing the informed consent form, or the date of signing the informed consent form still within 5 half-lives of the drug from the last dose in the last clinical trial (whichever is longer);
16. Patients with poor compliance due to physiological, family, social, geographic and other factors, and failure to follow the study protocol and the follow-up plan;
17. Patients with contraindications to cyclophosphamide, fludarabine, IL-2, or other drugs related to the study treatment;
18. Comorbidities requiring treatment with systemic corticosteroids (dexamethasone at a dose of ≥5 mg/day or other corticosteroids at the equivalent dose) or other immunosuppressive drugs within 12 weeks after the study treatment starts as judged by the investigator;
19. Women who are breastfeeding and are unwilling to stop breastfeeding;
20. Any other conditions that are, in the opinion of the investigator, not suitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | 4 weeks
  Proportion of patients with DLT
Adverse Events (AEs) | 96 weeks
  Incidence and severity of adverse events
Serious Adverse Events (SAEs) | 96 weeks
  Incidence and severity of serious adverse events

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 12 weeks
  The percentage of participants who achieved Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1
Disease Control Rate (DCR) | 12 weeks
  The percentage of participants who achieved Complete Response (CR) or Partial Response (PR) or Stable disease (SD) based on RECIST version 1.1
Changes in Serum Tumor Markers compared to Baseline | 12 weeks
  Changes of tumor markers in serum detected by immunofluorescence compared to baseline level, including carbohydrate antigen 19-9 (CA19-9), carcinoembryonic antigen (CEA), and carbohydrate antigen 12-5 (CA12-5)
Duration of response (DOR) | 96 weeks
  DOR is defined as the time from the first evaluation of a tumor as CR or PR to the first evaluation as PD or death from any cause
Time to response (TTR) | 96 weeks
  TTR is defined as the time between cell infusion and initial disease assessment as CR or PR
Progression-free survival (PFS) | 96 weeks
  PFS is defined as the time from the date of cell infusion until the date of tumor progression or death from any cause
Overall survival (OS) | 96 weeks
  OS is defined as the time between the date of cell infusion and the death of the patient for any reason
TCR gene copies | 96 weeks
  TCR gene copies detected by qPCR in peripheral blood
TCR-T cell counts | 96 weeks
  TCR-T cell counts detected by flow cytometry in peripheral blood
Proportion of patients with anti-IX001 antibodies in peripheral blood | 96 weeks
  Anti-drug Antibodies

CONTACTS AND LOCATIONS:
Overall Officials: MingHua Yu, Dr., Principal Investigator — Shanghai Pudong Hospital
Locations (1):
- Shanghai Pudong Hospital, Shanghai, Shanghai Municipality, China